CLINICAL TRIAL: NCT01413139
Title: 4-EVER Study - Physician-Initiated Trial Investigating the Safety of the Full 4F Endovascular Treatment Approach of Infra-Inguinal Arterial Stenotic Disease
Brief Title: 4-EVER : a Trial Investigating the Safety of 4F Endovascular Treatment of Infra-Inguinal Arterial Stenotic Disease
Acronym: 4-EVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-100701
Record Dates: First submitted 2010-07-01; First posted 2011-08-10 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Peripheral Vascular Disease; Claudication
Keywords: peripheral Vascular Disease; claudication; rest pain
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4F portfolio products from Biotronik (Other): The devices under investigation are the 4F portfolio products from Biotronik: Astron pulsar / Astron Pulsar-18, Fortress, Passeo-18 and Cruiser-18.
  Interventions: Device: 4F portfolio products from Biotronik

INTERVENTIONS:
Device: 4F portfolio products from Biotronik — 4F portfolio products from Biotronik: Astron pulsar / Astron Pulsar-18, Fortress, Passeo-18, Cruiser-18
  Other Names: Astron pulsar; Astron Pulsar-18; Fortress; Passeo-18; Cruiser-18

SUMMARY:
The objective of this clinical investigation is to evaluate puncture site complication rate as well as the short- and long-term (up to 24 months) outcome of treatment by means of Astron Pulsar / Astron Pulsar-18 stent implantation in symptomatic (Rutherford 2-4) femoro-popliteal arterial stenotic or occlusive lesions, using 4F compatible devices of BIOTRONIK and without the use of a closure device.

The hypothesis is that the primary patency at 12 months is non-inferior to the primary patency obtained in the Durability study (72.2%).

ELIGIBILITY:
Inclusion Criteria:

* De novo, restenotic or reoccluded lesion located in the femoropopliteal arteries suitable for endovascular treatment
* Patient presenting with a score from 2 to 4 according to the Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the predefined time intervals times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrollment in the study
* Prior to enrollment, the target lesion was crossed with standard guidewire manipulation
* Patient is eligible for treatment with 4F compatible devices

Angiographic Inclusion Criteria:

* The target lesions are located within the native superficial femoral artery: Distal point 3 cm above knee joint and 1 cm below the origin of the profunda femoralis.
* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion
* Length of the target lesion is =20 cm by visual estimation and can be covered with one stent
* Target vessel diameter visually estimated is =4 mm and =6.5 mm
* There is angiographic evidence of at least one-vessel-runoff to the foot

Exclusion Criteria:

* Presence of another stent in the target vessel that was placed during a previous procedure
* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
* Previous bypass surgery in the same limb
* Patients contraindicated for antiplatelet therapy, anticoagulants or thrombolytics
* Patients who exhibit persistent acute intraluminal thrombus at the target lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than 12 months
* Ipsilateral iliac artery treatment before target lesion treatment with a residual stenosis > 30%
* Use of thrombectomy, atherectomy or laser devices during procedure
* Any planned surgical intervention/procedure 30 days after the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not reached the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no reintervention | 12 months
  Primary patency at 12 months, defined as freedom from >50% restenosis

SECONDARY OUTCOMES:
Technical success | 1 day post-procedure
  Technical success, defined as the ability to cross and stent the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex imaging.
Puncture site complications | 10 days
  Number of puncture site complications in the absence of a closure device after intervention
Primary patency | 6- & 24-month follow-up
  Primary patency rate at 6- & 24-month follow-up, defined as freedom from >50% restenosis at 6 & 24 months as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no reintervention.
Clinical success | 6-, 12- & 24-month follow-up
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 6-, 12- & 24-month follow-up of one class or more as compared to the pre-procedure
Stent fracture rate at 12- & 24-month follow-up | 12- & 24-month follow-up
  Stent fracture rate at 12- & 24-month follow-up (in patient who were treated with stentplacement), as determined according the following classification on x-ray:
  1. Class 0 : no strut factures
  2. Class I : single tine fracture
  3. Class II : multiple tine factures
  4. Class III : Stent fracture(s) with preserved alignment of the components
  5. Class IV : Stent fracture(s) with mal-alignment of the components
  6. Class V : Stent fracture(s) in a trans-axial spiral configuration

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint Blasius, Dendermonde, Belgium
Locations (5):
- Belgium (3):
  - Imelda hospital, Bonheiden, Antwerpen
  - Universitair ziekenhuis antwerpen, Edegem, Antwerpen
  - AZ Sint Blasius, Dendermonde, Oost-Vlaanderen
- Germany (2):
  - Park-Krankenhaus Leipzig, Leipzig
  - St Fransiskus hospital, Münster

REFERENCES:
- [Derived] Bosiers M, Deloose K, Callaert J, Keirse K, Verbist J, Hendriks J, Lauwers P, D'Archambeau O, Scheinert D, Torsello G, Peeters P. 4-French-compatible endovascular material is safe and effective in the treatment of femoropopliteal occlusive disease: results of the 4-EVER trial. J Endovasc Ther. 2013 Dec;20(6):746-56. doi: 10.1583/13-4437MR.1. PMID 24325689